CLINICAL TRIAL: NCT00671684
Title: Endoscopic Mucosal Resection for the Diagnosis of a-Ganglionosis, a Controlled Prospective Trial
Brief Title: Endoscopic Mucosal Resection (EMR) for Diagnosis of Hirschsprung's Disease
Acronym: EDGE
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Leonel Rodriguez, MD, Massachusetts General Hosptial
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2007P001577
Record Dates: First submitted 2008-05-01; First posted 2008-05-05 (Estimated); Last update posted 2008-05-05 (Estimated); Status verified 2008-05

CONDITIONS: Chronic Constipation; Hirschsprung's Disease
Keywords: Hirschsprung's disease; Constipation; Endoscopy, digestive system; Diagnosis; Colonoscopy
MeSH Terms: conditions — Hirschsprung Disease; Constipation; Disease | interventions — Endoscopic Mucosal Resection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: Endoscopic Mucosal Resection (EMR) — EMR is a common procedure in gastroenterology. The technique involves placing a band around a piece of mucosa in the GI tract. The band and the tissue are then removed using a cautery snare. The technique can be used to obtain tissue for diagnostic purposes or to remove lesions for therapeutic purposes.

SUMMARY:
The purpose of this study is to compare the diagnostic yield with endoscopic mucosal resection (EMR) in hirschsprung's disease versus that of standard rectal suction biopsy. In order to compare EMR versus rectal suction biopsy, patients' diagnostic specimens will be analyzed by tissue size, the presence of submucosal tissue, and positive acteylcholinesterase staining. Additionally, the proportion of patients who would have required subsequent full thickness surgical biopsy with each technique will be compared. Biopsy results will be compared with clinical data including history, Bristol stool scale, anorectal manometry results and SITZ markers studies. Finally, the estimated costs that would have been incurred with each method will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Patients offered a rectal suction biopsy

Exclusion Criteria:

* any contraindication to general anesthesia or conscious sedation
* contraindication to endoscopy
* untreated or unmanageable coaguloapathy
* thrombocytopenia (<50)
* inability to provide informed consent.

Min Age: 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2007-10; Primary Completion 2009-04 (Estimated); Study Completion 2009-04 (Estimated)

PRIMARY OUTCOMES:
The major goal of this study is to test the hypothesis that EMR will result in a higher proportion of diagnostic specimens than RSB in patients sent for rectal suction biopsy. | April 2009

SECONDARY OUTCOMES:
Secondary outcome variables include the size of the specimen, the presence of ganglionic tissue, the presence of submucosal tissue, and the positivity of the acetylcholinesterase stain. | April 2009

CONTACTS AND LOCATIONS:
Overall Officials: Field F Willingham, MD, MPH, Study Director — MGH; Garrett C Zella, MD, Study Director — MGH; Mari Mino-Kenudson, MD, Study Director — MGH; Braden Kuo, MD, Principal Investigator — MGH; William R Brugge, MD, FASGE, Study Director — MGH; Leonel Rodriguez, MD, Principal Investigator — MGH; Clarissa Foy, NP, Study Director — MGH
Locations (1):
- Massachusetts General Hosptial, Boston, Massachusetts, United States